CLINICAL TRIAL: NCT02656706
Title: Adjuvant Nivolumab and Low Dose Ipilimumab for Stage III and Resected Stage IV Melanoma: A Phase II Brown University Oncology Research Group Trial
Brief Title: Adjuvant Nivolumab & Low Dose Ipilimumab for Stage III & Resected Stage IV Melanoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: Rhode Island Hospital (Other); The Miriam Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BrUOG 324
Record Dates: First submitted 2016-01-11; First posted 2016-01-15 (Estimated); Results first posted 2022-03-22 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2025-12

CONDITIONS: Melanoma
Keywords: Adjuvant melanoma; Advanced melanoma
MeSH Terms: conditions — Melanoma | interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Adjuvant treatment (Experimental): Ipilumumab:1mg/kg q6weeks (1 dose per cycle, 4 planned treatments over 6 months total) Nivolumab:3mg/kg q2weeks (3 doses per cycle, 12 planned treatments over 6 months total)
  Interventions: Drug: Ipilumumab; Drug: Nivolumab

INTERVENTIONS:
Drug: Ipilumumab
Drug: Nivolumab

SUMMARY:
Effective adjuvant treatment can increase cure in patients with high-risk resected melanoma. High dose interferon is a standard of care in the adjuvant setting but is highly toxic and marginally effective. The combination of ipilimumab and nivolumab is the most active regimen in patients with advanced melanoma so there is clear rationale to test this regimen in the adjuvant setting. Investigators are testing if nivolumab 3mg/kg every 2 weeks with 1mg/kg ipilimumab every 6 weeks in the high risk adjuvant setting. The duration of therapy will be six months.

DETAILED DESCRIPTION:
See above summary

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically proven melanoma. The primary site of melanoma may be cutaneous on other body site such as ocular or anorectal. Documentation required to be sent to BrUOG.
* Completely resected stage III (lymph node positive) or resected stage IV disease. Patients with stage T4BN0 are also eligible. It is required that patients with stage IIIA disease have > 1mm nodal involvement via pathology assessment of the resected node. All patients must be disease free to be eligible.
* No prior treatment for melanoma other than surgical resection or radiation. At least 4 weeks since prior surgery and 3 weeks since prior radiation to registration date.
* Age >/= 18 years
* ECOG performance status 0-1
* Patients must have organ and marrow function as defined below within 14 days of study entry:

Hematologic Absolute neutrophil count (ANC) >/= 1.5 X 109/L; Hemoglobin >/= 9.5 g/dL; Platelets >/= 100 X 109/L; Total Bilirubin ≤ 1.5 x ULN except subjects with normal direct bilirubin or those with known Gilbert's syndrome. Send information to BrUOG if patient has known Gilbert's syndrome AST and ALT </= 2.5 X ULN Albumin >/= 2.5 g/dL Renal Creatinine OR Calculated creatinine clearance : Creatinine </= 1.5 mg/dl or creatinine clearance > 50ml/min

* No clinically significant coagulation disorder as defined by the treating MD. Therapeutic use of anticoagulants is permissible. Add to concomitant medication log if applicable.
* Not pregnant and not nursing. Women of child bearing potential must have a negative serum pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 7 days prior to Day 1 of treatment. Post-menopausal women (surgical menopause or lack of menses >12 months) do not need to have a pregnancy test, please document status.
* Confirmation of informed consent.
* Men and women of childbearing potential enrolled in this study must agree to use adequate barrier birth control measures during the course of the study and up to 2 months after end of treatment.

Exclusion Criteria:

* Currently receiving cancer therapy (chemotherapy, radiation therapy, immunotherapy, or biologic therapy) or investigational anti-cancer drug
* Brain metastases, whether resected or not, and any known leptomeningeal disease or known bone metastases.
* Pregnant or breastfeeding female
* Unwillingness or inability to follow the procedures required in the protocol, to document
* Any serious or uncontrolled medical disorder that, in the opinion of the investigator, may increase the risk associated with study participation or study drug administration, impair the ability of the subject to receive protocol therapy, or interfere with the interpretation of study results.
* Prior malignancy active within the previous 2 years except for locally curable cancers that have been apparently cured, such as basal or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the prostate, cervix, or breast. Documentation required to be sent to BrUOG
* Subjects with active, known or suspected autoimmune disease. Subjects with vitiligo, controlled type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll.
* Subjects with a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids and adrenal replacement doses >10mg daily of prednisone equivalents are permitted in the absence of active autoimmune disease.
* Prior treatment with an anti-PD-1, anti-PD-L1 or anti-CTLA-4 antibody
* Any positive test result for hepatitis B or C virus indicating acute or chronic infection
* Known history of testing positive for human immunodeficiency virus or known acquired immunodeficiency syndrome
* History of severe hypersensitivity reaction to any monoclonal antibody.
* Patients with unstable angina (anginal symptoms at rest) or new-onset angina (began within the last 3 months) or myocardial infarction within the past 6 months.
* History of autologous transplant or organ allograft even if not taking immunosuppressive medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2019-03 (Actual); Study Completion 2026-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Howard Safran, MD, Study Chair — BrUOG Study Chair
Locations (1):
- Rhode Island Hospital and The Miriam Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Adjuvant Treatment
Started | 22
Completed | 21
Not Completed | 1
Not completed — Insurance Denial | 1

BASELINE CHARACTERISTICS:
Arm/Group | Adjuvant Treatment
Number analyzed (Participants) | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 9
Age, Continuous [Mean (Full Range); unit: years] | 57 [25 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 21
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 21

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Related Toxicities
Time Frame: From day 1 of treatment through 30 days post the last dose of drug, for a total of about 7 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Adjuvant Treatment
Number analyzed (Participants) | 21
Participants | 21

2. Primary Outcome: Number of Participants With Progression-free and Survival Overall
Time Frame: Post treatment for up to 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Adjuvant Treatment
Number analyzed (Participants) | 21
Participants
  2-year progression free survival | 18
  2-year overall survall | 19

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time a signed and dated ICF is obtained until 30 days after the last dose of treatment, or until the subject withdrew consent from study participation, whichever occurs first. All cause mortality was assessed from the time a signed and dated ICF is obtained until up to 5 years post treatment (approximately 5.5 years).
Arm/Group | Adjuvant Treatment
All-Cause Mortality (participants affected / at risk) | 2/21
Serious Adverse Events (participants affected / at risk) | 11/21
Other Adverse Events (participants affected / at risk) | 20/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Adjuvant Treatment (N=21)
Cardiac Disorders, other (Cardiac disorders) | 1 — Unstable angina
Pericardial effusion (Cardiac disorders) | 1
Adrenal insufficiency (Endocrine disorders) | 1
Endocrine disorders, other (Endocrine disorders) | 1
Colitis (Gastrointestinal disorders) | 2
Diarrhea (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Vomitting (Gastrointestinal disorders) | 1
Pain (General disorders) | 2
Immune system disorders, other (Immune system disorders) | 3 — Immune Mediated Hepatitis
Infection (Infections and infestations) | 1
Alanine aminotransferase increased (Investigations) | 1
Creatinine increased (Investigations) | 2
Dehydration (Metabolism and nutrition disorders) | 3
Hyperglycemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Meningismus (Nervous system disorders) | 1
Stroke (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Confusion (Psychiatric disorders) | 1
Chylothorax (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Adjuvant Treatment (N=21)
Anemia (Blood and lymphatic system disorders) | 10
Adrenal insufficiency (Endocrine disorders) | 2
Hyperthyroidism (Endocrine disorders) | 7
Hypothyroidism (Endocrine disorders) | 2
Blurred vision (Eye disorders) | 5
Colitis (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 2
Diarrhea (Gastrointestinal disorders) | 8
Dry mouth (Gastrointestinal disorders) | 4
Gastroesophageal reflux disease (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 11
Vomiting (Gastrointestinal disorders) | 4
Edema (General disorders) | 6
Fatigue (General disorders) | 13
Non cardiac chest pain (General disorders) | 3
Pain (General disorders) | 9
Immune system disorders, other (Immune system disorders) | 2
Immune system disorders, other (Immune system disorders) | 2 — Immune mediated hepatitis
Infection (Infections and infestations) | 6
Alanine aminotransferase increased (Investigations) | 8
Aspartate aminotransferase increased (Investigations) | 6
Blood bilirubin increased (Investigations) | 3
Creatinine increased (Investigations) | 4
Hemoglobin increased (Investigations) | 5
Lymphocyte count decreased (Investigations) | 9
Platelet count decreased (Investigations) | 5
Weight gain (Investigations) | 3
Weight loss (Investigations) | 6
Anorexia (Metabolism and nutrition disorders) | 3
Dehydration (Metabolism and nutrition disorders) | 4
Hyperglycemia (Metabolism and nutrition disorders) | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 4
Hypocalcemia (Metabolism and nutrition disorders) | 4
Hypokalemia (Metabolism and nutrition disorders) | 13
Hypomagnesemia (Metabolism and nutrition disorders) | 9
Hyponatremia (Metabolism and nutrition disorders) | 12
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Paresthesia (Nervous system disorders) | 2
Anxiety (Psychiatric disorders) | 4
Insomnia (Psychiatric disorders) | 6
Acute kidney injury (Renal and urinary disorders) | 2
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 3
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2
Pruritus (Skin and subcutaneous tissue disorders) | 8
Rash (Skin and subcutaneous tissue disorders) | 10
Skin and subcutaneous tissue disorders, other (Skin and subcutaneous tissue disorders) | 2 — Pimple axilla
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2018-12-08): https://cdn.clinicaltrials.gov/large-docs/06/NCT02656706/Prot_SAP_ICF_000.pdf